CLINICAL TRIAL: NCT05710588
Title: The Effectiveness of Motor-motor and Motor-cognitive Dual-task Training Interventions on Balance in People With Parkinson's Disease: a Feasibility Study of a Randomized Clinical Trial
Brief Title: The Effectiveness of Motor-motor and Motor-cognitive Dual-task Training Interventions on Balance in People With Parkinson's Disease: a Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Nesibe Cakmak, Principal Investigator, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3332
Record Dates: First submitted 2022-12-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; balance; dual-task training; home-based training; feasibility; acceptability
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: There are two different intervention groups: M-DTT and C-DTT. Participants will be allocated to either M-DTT or C-DTT group.
Who Masked: Participant
Masking Description: Participants will know they are allocated to one group randomly but they will not know which group is this.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-DTT group (Experimental): This group has motor-motor dual task training-balance related tasks as primary task (e.g. marching, stepping) and motor tasks as secondary task (e.g. touching wall, popping a fidget toy).
  Interventions: Other: motor-motor dual-task training
- C-DTT group (Experimental): This group has motor-cognitive dual-task training-balance related tasks as primary task (e.g. marching, stepping) and cognitive tasks as secondary task (e.g. repeating tongue twisters, counting backwards from 100).
  Interventions: Other: motor-cognitive dual-task training

INTERVENTIONS:
Other: motor-motor dual-task training — The intervention compromises balance-related tasks which are selected among the tasks often used in balance rehabilitation and motor secondary tasks might be required hand dexterity like popping a fidget toy or reaching ability like touching wall. All sessions will be individual. The initial training session will be undertaken in University of Plymouth. This will be followed by a recorded training video programme which can be accessible through Panopto- a University-led, web-based platform- undertaken in the participants' home for 30 minute sessions, three times a week over 6 weeks.
  Arms: M-DTT group
Other: motor-cognitive dual-task training — The intervention compromises (1) balance-related tasks which are selected among the tasks often used in balance rehabilitation and (2) cognitive secondary tasks might required to activate sensory and cognitive systems like listening podcast and memorizing the details about it or reading a tongue twister and repeating. intervention delivery will be the same with M-DTT group.
  Arms: C-DTT group

SUMMARY:
This study aims to test the feasibility and acceptability of home-based motor-motor dual-task training and motor-cognitive dual-task training interventions, and balance-related outcome measures which may be used in an anticipated future randomized control trial intended to determine the superiority of these dual-task training interventions.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a complex, progressive neurodegenerative disorder characterized by the degeneration of dopaminergic neurons in the basal ganglia. Balance impairment is one of the major problems in people with PD, often manifested at a stage of mild to moderate disease severity.

Balance impairments in people with PD affect different domains of balance control: (1) postural sway during quiet stance, (2) automatic postural responses to external perturbations, (3) anticipatory postural adjustment, such as is seen before gait initiation (APAs), and (4) dynamic balance during walking. Therefore, it is important to focus on upright, bipedal balance in people with PD.

Physiotherapy approaches have found to be effective in improving balance-related motor impairments in people with PD. Dual-task training is one of these physiotherapy approaches. This involves simultaneous performance of a primary task and a second discrete task which is independent from the primary task. The primary task is usually a motor task like standing or walking, and the secondary task is either a motor task or a cognitive task such as carrying an object or talking. Dual-task training (DTT) has demonstrated to be effective in enhancing balance control and promoting interactions between the motor and cognitive systems. Two systematic reviews have been undertaken in this area. One found DTT improved balance in people with mild to moderate PD. The second included a meta-analysis, reporting a moderate effect in favor of DTT group on functional balance. However, there remains a lack of evidence about the superiority of motor-motor dual-task training (M-DTT) versus motor-cognitive dual-task training (C-DTT) in terms of improving balance.

A scoping review which is a part of this project shows that only one study compares the effectiveness of M-DTT and C-DTT on balance but this study has some methodological limitations. So, there is a need for a future randomized control trial to investigate the superiority of M-DTT and C-DTT on balance in people with PD.

The COVID-19 pandemic has shifted physiotherapy deliveries to telerehabilitation . A recent systematic review showed that telerehabilitation is feasible for people with PD and effective in improving and/or maintaining balance and gait and some non-motor aspects (quality of life, patient satisfaction) of the disease. So, DTT delivered to people in their homes via telerehabilitation may be an applicable alternative to traditional face-to-face physiotherapy service delivery.

The scoping review showed that there is some published evidence about home-based DTT, but no studies have investigated and compared the effectiveness of M-DTT and C-DTT interventions on balance in people with mild-moderate PD. For instance, one case study used C-DTT as a part of exergaming plus treadmill intervention in a home setting, but they only applied C-DTT, and there was no other type of DTT as a comparison in their study.

So, this study aims to test the feasibility and acceptability of the M-DTT and C-DTT interventions, and balance-related outcome measures which may be used in an anticipated future randomized control study intended to determine the superiority of these dual-task training interventions.

Study Objectives:

* To test the feasibility and acceptability of home-based C-DTT and M-DTT interventions.
* To assess the acceptability and utility of the outcome measures, from the participant perspective.
* To assess safety by monitoring for any adverse events or serious adverse events.
* To assess the feasibility and acceptability of the safety monitoring process, from the participant perspective.
* To assess the potential effect of C-DTT and M-DTT on standing and walking balance.

ELIGIBILITY:
Inclusion Criteria:

* Self-report a diagnosis of PD
* Are categorized as having mild to moderate PD (based on scoring of the modified UPDRS scale, undertaken via an online interview).
* Can understand and follow instructions.
* Can independently, or with help of a supporter, complete self-report outcome measures.
* Can use web-based/online applications independently, or with help of a supporter.
* Have a supporter (carer, spouse, family member aged ≥18) who is willing and able to act as an exercise buddy.
* Have an available safe training area according to the definition: A 2 meter square clear area immediately next to a wall, with no trip hazards and with the potential to place a chair within the space (for seated rests). The wall needs to be free from hanging objects or shelves and not wallpapered or featuring flaking plaster. This is to ensure safety during training and prevent unintended damage to the wall. (Closed doors may be considered as part of the 'wall' only if they can be securely shut, so that should a near-fall occur with participant's falling against the door, they would not open. They should also be guaranteed not to be opened by other household members (including pets) during the training session (which could potentially cause a fall)).

Exclusion Criteria:

* Neurological, orthopaedic or any other current medical problems other than PD which can affect standing balance (such as stroke, cerebellar disorders, a vestibular impairment, a skeletal fracture (occurred within past six months), severe visual impairment) as this could both risk safety within a standardized training protocol and independently affect treatment outcomes.
* Severe deafness without the support of a signing translator, to ensure that participants will be able to effectively receive communication.
* Those unable to communicate in English, as no translation will be available, and communication is essential in ensuring safety.
* Unable to stand independently for more than 1 minute without requiring external postural support, to ensure safety (and prevent falls) during training and outcome measurement.
* Unsuitable training area according to the definition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
change from baseline body sway at 6 weeks | Measurements will be conducted at baseline and after the 6-weeks training programme.
  body sway will be recorded for mediolateral (ML) and anteroposterior (AP) directions. A sensor will calculate the orientation euler angles (XYZ Earth fixed type) in degrees. Measurements will be standing 45 sec in comfortable position-eyes open, comfortable position-eyes closed, and feet are in 4 cm apart-eyes open on firm surface.
change from baseline MiniBESTest score at 6 weeks | Measurements will be conducted at baseline and after the 6-weeks training programme. Higher scores represent better outcome
  standing and functional balance assessment
Acceptability questionnaire | at the end of week 2 of the training programme.
  Participants' perception regarding the intervention (individual task difficulty, progression, satisfaction, enjoyment, etc.), will be asked via an online 5-point Likert scale questionnaire.
Acceptability questionnaire | at the end of week 4 of the training programme.
  Participants' perception regarding the intervention (individual task difficulty, progression, satisfaction, enjoyment, etc.), will be asked via an online 5-point Likert scale questionnaire.
Acceptability questionnaire | at the end of week 6 of the training programme.
  Participants' perception regarding the intervention (individual task difficulty, progression, satisfaction, enjoyment, etc.), will be asked via an online 5-point Likert scale questionnaire.
the number of total hours of undertaken training sessions over 6 weeks training programme | at the end of the 6 weeks training programme
  Panopto (University of Plymouth licensed online video streaming platform) enables to record participants adherence and attendance rates to the training sessions. the number of hours watched will be recorded for each session and for 6 weeks training programme in total.
semi-structured interviews | a week after completion of the training programme
  to assess acceptability their perception regarding outcome measures (trustfulness, etc.), monitoring (e.g. difficulty, independence, etc.), and overall intervention will be asked in an online semi-structured interviews.
safety assessment by monitoring for any adverse events | at the end of the 6 weeks training programme.
  for safety assessment the number of falls and near falls (stumbling/losing balance not resulting with a fall) during the training programme will be recorded within training workbook by participants. Semi-structured interviews will allow to understand how those falls/near falls occured. Also, any serious adverse events that resulted any injuries will be asked during this interviews.

OTHER OUTCOMES:
Demographic and medical information form | At baseline
  Age, gender, number of years after diagnosis, working status, other medical conditions, the number of falls in last month.
self-report MDS-UPDRS-II questionnaire | At baseline
  This questionnaire asks questions how Parkinson's affects patients' experiences of daily life to understand their disease severity. Higher scores represent higher severity.
Mini Mental State Examination Test | At baseline
  A test of cognitive function. Higher scores represent better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bunn, Study Director — University of Plymouth
Locations (1):
- University of Plymouth, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The information from participants and all collected and processed data will be used only for the purpose of this study by the research team. University of Plymouth will keep data about participants for 10 years after the study has finished and then will destroy the data permanently.

REFERENCES:
- [Background] De Freitas TB MS, PT, Leite PHW BS, Dona F PhD, PT, Pompeu JE PhD, PT, Swarowsky A PhD, PT, Torriani-Pasin C PhD, PT. The effects of dual task gait and balance training in Parkinson's disease: a systematic review. Physiother Theory Pract. 2020 Oct;36(10):1088-1096. doi: 10.1080/09593985.2018.1551455. Epub 2018 Dec 3. PMID 30501424
- [Background] Hasegawa N, Shah VV, Harker G, Carlson-Kuhta P, Nutt JG, Lapidus JA, Jung SH, Barlow N, King LA, Horak FB, Mancini M. Responsiveness of Objective vs. Clinical Balance Domain Outcomes for Exercise Intervention in Parkinson's Disease. Front Neurol. 2020 Sep 25;11:940. doi: 10.3389/fneur.2020.00940. eCollection 2020. PMID 33101161
- [Background] Li Z, Wang T, Liu H, Jiang Y, Wang Z, Zhuang J. Dual-task training on gait, motor symptoms, and balance in patients with Parkinson's disease: a systematic review and meta-analysis. Clin Rehabil. 2020 Nov;34(11):1355-1367. doi: 10.1177/0269215520941142. Epub 2020 Jul 13. PMID 32660265
- [Background] Pourkhani, T., Daneshmandi, H., Norasteh, A., Bakhshayesh Eghbali, B. & Sedaghati, P. (2019) 'The Effect of Cognitive and Motor Dual-Task Training on Improvement of Balance and Some Spatiotemporal Gait Parameters in People With Idiopathic Parkinson Disease.'. Caspian J Neurol Sci., 5 (4), pp. 190-198.
- [Background] Radder DLM, Ligia Silva de Lima A, Domingos J, Keus SHJ, van Nimwegen M, Bloem BR, de Vries NM. Physiotherapy in Parkinson's Disease: A Meta-Analysis of Present Treatment Modalities. Neurorehabil Neural Repair. 2020 Oct;34(10):871-880. doi: 10.1177/1545968320952799. Epub 2020 Sep 11. PMID 32917125
- [Background] Vallabhajosula S, McMillion AK, Freund JE. The effects of exergaming and treadmill training on gait, balance, and cognition in a person with Parkinson's disease: A case study. Physiother Theory Pract. 2017 Dec;33(12):920-931. doi: 10.1080/09593985.2017.1359867. Epub 2017 Aug 16. PMID 28812419
- [Background] Vellata C, Belli S, Balsamo F, Giordano A, Colombo R, Maggioni G. Effectiveness of Telerehabilitation on Motor Impairments, Non-motor Symptoms and Compliance in Patients With Parkinson's Disease: A Systematic Review. Front Neurol. 2021 Aug 26;12:627999. doi: 10.3389/fneur.2021.627999. eCollection 2021. PMID 34512495